CLINICAL TRIAL: NCT07197359
Title: Detecting Asymmetry With Artificial Intelligence: Consistency Evaluation of the Looksmaxxing Application in Photo-Based Facial Analysis
Brief Title: Looksmaxxing AI for Chin Deviation Detection
Status: Active, not recruiting | Type: Observational
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Seda Sağoğlu, Research assistant, Konya Necmettin Erbakan Üniversitesi
Other Study IDs: 2025/635
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Mandibular Asymmetry
Keywords: chin asymmetry; photographic analysis; artificial intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Chin Deviation: Participants clinically diagnosed with chin deviation (laterognathia) based on frontal facial examination.
  Interventions: Other: Looksmaxxing AI Facial Analysis
- Without Chin Deviation: Participants with clinically normal chin position confirmed by frontal facial examination.
  Interventions: Other: Looksmaxxing AI Facial Analysis

INTERVENTIONS:
Other: Looksmaxxing AI Facial Analysis — Participants' standardized frontal facial photographs will be analyzed using the Looksmaxxing AI application (versions 4o and 5) to determine the presence or absence of chin deviation relative to the facial midline.

SUMMARY:
This study aims to evaluate whether an artificial intelligence application called Looksmaxxing AI will be able to correctly identify chin deviation (chin asymmetry) from standard frontal facial photographs. A total of 540 photographs will be included in the study. The eye areas will be covered to protect identity. Each photo will be analyzed by the AI, and its answers will be compared with clinical reality. The accuracy of two versions of the software (Looksmaxxing 4o and 5) will be assessed. The results may help show whether simple photo-based analysis can support early detection of chin asymmetry, especially in areas with limited access to orthodontic examination.

DETAILED DESCRIPTION:
This observational study will investigate the accuracy of the Looksmaxxing AI application in detecting chin deviation based on standardized frontal facial photographs. A total of 540 images will be included. To protect identity, the eye areas of all participants will be covered. The AI will be asked to determine whether chin deviation is present relative to the midline of the face (excluding the nose).

The study population will consist of two equally sized groups:

270 individuals with clinically observed chin deviation (laterognathia)

270 individuals with clinically normal chin position

The responses provided by Looksmaxxing AI will be compared with the clinical reality and recorded for accuracy. Both versions of the software, Looksmaxxing 4o and Looksmaxxing 5, will be analyzed to evaluate their level of consistency with clinical findings. Results will be reported as accuracy percentages. In addition, prediction accuracy will be compared between individuals with and without chin deviation, and the statistical significance of the difference will be tested using the Chi-square method.

ELIGIBILITY:
Inclusion Criteria:

* Absence of any craniofacial anomaly

No major wound or scar in the facial or neck region

No history of previous orthodontic treatment

For male participants: absence of a long beard that could affect the appearance of the chin

Availability of standardized frontal facial photographs taken in natural head position

Exclusion Criteria:

* Photographs in which the patient's face appears slightly angled or turned sideways

Blurred or low-quality photographs with reduced clarity

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Standardized frontal facial photographs of 90 individuals (540 images in total) will be analyzed. The study population consists of two equal groups: 270 photographs from individuals with clinically observed chin deviation (laterognathia) and 270 photographs from individuals with clinically normal chin position.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Looksmaxxing AI in Detecting Chin Deviation | At study completion (October 2025)
  The proportion of correct classifications (presence or absence of chin deviation) made by the Looksmaxxing AI application compared to the clinical gold standard, expressed as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (facial photographs) will not be shared due to privacy concerns and the risk of re-identification. Only aggregated and anonymized results will be published.

REFERENCES:
- See also: This article reports the use of deep learning for automatic classification of orthodontic photographs, providing methodological background relevant to AI-based facial asymmetry detection. — https://bmcoralhealth.biomedcentral.com/articles/10.1186/s12903-022-02466-x